CLINICAL TRIAL: NCT04963465
Title: Assessing the Accuracy of Amniotic Fluid Ferning in the Second Trimester in the Diagnosis of Preterm Prelabor Rupture of Membranes
Brief Title: The Accuracy of Amniotic Fluid Ferning in the Second Trimester in the Diagnosis of Preterm Prelabor Rupture of Membranes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Albany Medical College (Other)
Responsible Party: Sponsor
Other Study IDs: 6229
Record Dates: First submitted 2021-07-06; First posted 2021-07-15 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Preterm Premature Rupture of Membrane; Amniotic Fluid Leakage
MeSH Terms: conditions — Preterm Premature Rupture of the Membranes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Before rupture of membranes: Vaginal swab collection prior to iatrogenic rupture of membranes
  Interventions: Diagnostic Test: Ferning on microscopy
- After rupture of membranes: Vaginal swab collection after iatrogenic rupture of membranes
  Interventions: Diagnostic Test: Ferning on microscopy

INTERVENTIONS:
Diagnostic Test: Ferning on microscopy — Amniotic fluid ferning will be assessed in the cohort before known rupture of membranes and after known rupture of membranes

SUMMARY:
Although much investigation has been done on the use of ferning in the second and third trimesters, particularly with the development of rapid protein clinical assays, there appears to be lower ferning rates in clinical practice with traditional techniques compared to previous published research on the subject. Much of the older study designs are lacking in detail and lack a large enough sample sizes at each gestational age to appropriately interpret the significance of ferning results by gestational age. Additionally, a large premise for the current tests used to diagnose rupture of membranes is based on these older studies. Given this, we propose collecting amniotic fluid vaginally to evaluate for the presence of ferning in the second trimester to determine if there is a difference in ferning based on gestational age as well as the time interval after rupture of membranes in which ferning can observed on microscope examination.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* English speaking
* singleton or multi fetal gestation
* between 15 and 24 weeks gestation
* undergoing elective pregnancy termination

Exclusion Criteria:

* known rupture of membranes or anhydramnios

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective observational study including pregnant women 18 years or older who present for pregnancy termination, between 15 and 24 weeks gestation. Women with a singleton or multi-fetal gestation, who have previously established dating based on a first trimester ultrasound or ultrasound prior to 22 weeks gestation, will be included. Exclusion criterion are women who are less than 18 years of age, non-English speaking, and rupture of membranes or anhydramnios (no measurable amniotic fluid on ultrasound) at the time of data collection in the operating room.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-09-17 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Ferning | 1 minute
  the presence of amniotic fluid ferning
Ferning | 5 minutes
  the presence of amniotic fluid ferning
Ferning | 10 minutes
  the presence of amniotic fluid ferning
Ferning | 15 minutes
  the presence of amniotic fluid ferning
Ferning | 20 minutes
  the presence of amniotic fluid ferning

CONTACTS AND LOCATIONS:
Overall Officials: OBGYN Research Director, Principal Investigator — Albany Medical College
Locations (1):
- Albany Medical Center, Albany, New York, United States

IPD SHARING:
Plan to Share IPD: No